CLINICAL TRIAL: NCT01301781
Title: A Pilot Efficacy Evaluation of BLI801 Laxative in Constipated Adults
Brief Title: BLI801 Laxative in Constipated Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLI801-201
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BLI801 laxative (Experimental): BLI801 laxative - oral solution
  Interventions: Drug: BLI801
- Placebo (Placebo Comparator): BLI801 placebo - oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLI801 — BLI801 laxative - oral solution
  Arms: BLI801 laxative
Drug: Placebo — BLI801 placebo - oral solution
  Arms: Placebo

SUMMARY:
A pilot study to evaluate the safety and efficacy of BLI801 vs. placebo in constipated adults.

ELIGIBILITY:
Inclusion Criteria:

* Constipated, defined by ROME III definition
* Subject has < 3 satisfactory BMs during the run-in period

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon
* Subjects taking laxatives or prokinetic agents that refuse to discontinue these treatments.
* Subjects who are allergic to any BLI801 component
* Subjects taking narcotic analgesics or other medications known to cause constipation.
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures
* Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
* Subjects with an active history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
percentage of patients experiencing a bowel movement within 3 hours of the first study medication dose | 3 hours

SECONDARY OUTCOMES:
percentage of patients experiencing a complete/satisfactory bowel movement (BM) within 3 hours of first dose | 3 hours
serum chemistry | 7 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Advanced Clinical Research Institute, Anaheim, California
  - Jupiter Research, Jupiter, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - Long Island GI Research Group, Great Neck, New York